CLINICAL TRIAL: NCT06850324
Title: A Proof of Concept Study to Evaluate the Precision of ABL-101 Perfluorocarbon and Fluorine-19 Magnetic Resonance Imaging in Mapping of Atherosclerotic Plaque Composition and Inflammation in Patients Undergoing Carotid Endarterectomy
Brief Title: Evaluate the Precision of ABL-101 Perfluorocarbon and Fluorine-19 MRI for the Mapping of Atherosclerotic Plaque Composition and Inflammation in Patients Undergoing Carotid Endarterectomy
Acronym: PARFUME
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruud van Heeswijk (Other)
Responsible Party: Sponsor-Investigator, Ruud van Heeswijk, Dr PD MER1, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-113
Record Dates: First submitted 2025-02-24; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Atherosclerotic Disease, Carotid; Carotid Endarterectomy
Keywords: Mapping of Atherosclerotic Plaque Composition and Inflammation; Carotid Endarterectomy; ABL-101 Perfluorocarbon; Fluorine-19 Magnetic Resonance Imaging
MeSH Terms: conditions — Carotid Artery Diseases; Inflammation | interventions — Weights and Measures

STUDY DESIGN:
Intervention Model Description: Open label proof-of-concept phase II study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The perfluorocarbon tracer ABL-101 is infused as a single dosage of 3 mL/kg body weight (Experimental): The doses of ABL-101 is administered using an IV infusion pump in the arm at 3mL/kg body weight (to a notional maximum of 100kg, rounded to the nearest ml), at the rate of 15 mL/min (900ml/hour).
  Patients will undergo a 1 hour-imaging with 19F MRI, 16h-36h after end of PFC infusion.
  Interventions: Drug: ABL-101 is administered at 3mL/kg body weight (to a notional maximum of 100kg, rounded to the nearest ml), at the rate of 15 mL/min (900ml/hour).

INTERVENTIONS:
Drug: ABL-101 is administered at 3mL/kg body weight (to a notional maximum of 100kg, rounded to the nearest ml), at the rate of 15 mL/min (900ml/hour). — The doses of ABL-101 is administered using an IV infusion pump in the arm at 3mL/kg body weight (to a notional maximum of 100kg, rounded to the nearest ml), at the rate of 15 mL/min (900ml/hour). Patients will undergo a 1 hour-imaging with 19F MRI, 16h-36h after end of PFC infusion.

SUMMARY:
This study is aimed at patients suffering from carotid atherosclerosis. In the presence of atherosclerosis of the carotid arteries, one of the treatments that can be proposed is carotid endarterectomy, the aim of which is to remove the atherosclerotic plaque that obstructs the carotid artery and therefore increases the risk of developing a stroke. The risk of rupture of these plaques is primarily assessed by anatomical medical imaging: the degree of stenosis (narrowing) that the plaque causes most often informs the decision whether or not to proceed with surgery. However, it is well established that the degree of stenosis is not a very precise decision criterion: some plaques would never have ruptured, while others have ruptured even though no surgical intervention had been performed. It has since been discovered that the degree of inflammation is a much more accurate predictor of future rupture, but there is currently no reliable non-invasive imaging marker to measure plaque inflammation.

In this study, the investigators therefore evaluate a new marker, the perfluorocarbon ABL-101, for non-invasive imaging of inflammation in atherosclerotic plaque. To assess the marker's effectiveness in quantifying inflammation in plaque, the plaque will be analyzed microscopically after removal to obtain a more accurate measure of the degree of inflammation. This will enable us to assess the effectiveness of the non-invasive marker injection method versus the more invasive microscopic analysis of the removed plaque.

ABL-101 consists of a perfluorocarbon (PFC) emulsion, a liquid mixture in which PFC particles are dispersed. PFCs are chemical compounds containing only carbon and fluorine, and are known for their ability to transport large quantities of oxygen. Totally inert, PFCs cannot be broken down by the body and are eliminated naturally. Due to their small size, these particles are also captured by certain immune system cells and, combined with 19F-MRI, constitute a marker of inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent signed by the patient if capable of discernment or by the legally authorized representative if the patient is considered non capable of discernment or authorisation received from independent physician,
2. Age ≥ 18 years old,
3. Symptomatic atherosclerotic stenosis of the internal carotid artery ≥ 50% or asymptomatic atherosclerotic stenosis of the internal carotid artery ≥ 60% confirmed on at least two non-invasive imaging studies (Doppler, CT angiography, or MR angiography),
4. Planned for an elective or semi-urgent carotid endarterectomy (CEA) in 2 days at the earliest based on the current institutional and international guidelines.

Exclusion Criteria:

1. Known thrombocytopenia (platelet count <150x109/L) or history of platelet function disorder,
2. MRI with gadolinium-based contrast agents within 24 hours of the MRI scan of this trial,
3. Known allergy to ABL-101 or any of its constituents (including egg phospholipids),
4. Known current infection,
5. Any current medical condition causing impaired immunity (e.g. HIV infection, hyposplenism) or use of systemic immunosuppressant medication except for inhaled, nasal intra-articular or topical corticosteroids) on an ongoing basis or within the preceding 30 days,
6. Women who are pregnant or breast feeding,
7. Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, advanced cardiac failure, etc.), Known or suspected non-compliance, drug or alcohol abuse,
8. Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.,
9. Participation in another study with investigational drug within the 30 days preceding and during the present study,
10. Previous enrolment into the current study,
11. Enrolment of the investigator, his/her family members, employees and other dependent persons,
12. Inability to undergo MR imaging (e.g. incompatible implants, claustrophobia, etc.),
13. Any incapacitated patient that is not expected to recover to a point where they will personally be capable of discernment and able to provide informed consent.
14. A priori refusal to receive information concerning fortuitous discoveries which may contribute to the prevention, diagnosis and treatment of the disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between 19F MRI signal measured in the carotid plaque to be excised and CD45+ leukocytes number per mm2 in the excised plaque | The timepoint for primary outcome is the day of 19F MRI.
  The primary outcome of this study is the correlation between:
  * The average of 19F MRI signal measured in the carotid plaque to be excised, and
  * The average of CD45+ leukocytes number per mm2 in the excised plaque

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes